CLINICAL TRIAL: NCT01256437
Title: Double Blind Placebo Controlled Trial, for Evaluating Preventive Therapy With Either Oint Threolone Versus Synthomycine Versus Aqua Cream, for EGFR'I Induced Acneiform Rash
Brief Title: Evaluating Preventive Therapy With Oint Threolone, Synthomycine or Aqua Cream, for EGFR'I Induced Acneiform Rash
Acronym: EGFR'I
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, iris amitay, Iris Amitay-Laish, MD, Rabin Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 6046
Record Dates: First submitted 2010-12-07; First posted 2010-12-08 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Acneiform Rash
Keywords: Acneiform eruption; papulopustular; EGFR; cetuximab; erlotinib; gefitinib; panitumumab; eruption secondary to treatment with either cetuximab
MeSH Terms: conditions — Acneiform Eruptions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- ointment Threolone (Experimental): Treatment with topical application of combined anti inflammatory and anti bacterial agent.
  Interventions: Drug: Threolone ointment; Drug: ointment Synthomycine; Drug: Aqua cream
- ointment Synthomycine (Active Comparator): ointment once daily for 1 month
  Interventions: Drug: ointment Synthomycine; Drug: Aqua cream
- Aqua cream (Placebo Comparator)
  Interventions: Drug: Aqua cream

INTERVENTIONS:
Drug: Threolone ointment — ointment once daily for 1 month
  Arms: ointment Threolone
Drug: ointment Synthomycine — ointment once daily for 1 month
  Arms: ointment Synthomycine; ointment Threolone
Drug: Aqua cream — ointment once daily for 1 month

SUMMARY:
The investigators hypothesized that topical anti-inflammatory treatment could counteract the inflammatory reaction induced by EGFR'Is.

DETAILED DESCRIPTION:
The investigators hypothesized that topical anti-inflammatory treatment could counteract the inflammatory reaction induced by EGFR'Is.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are planed to initiate treatment with either cetuximab , erlotinib, gefitinib or panitumumab.

Exclusion Criteria:

* Patients who received any facial topical treatment / systemic antibiotics or any anti-inflammatory drug during the 2 weeks prior to study initiation.
* Known hypersensitivity to ointment Synthomycine or to Threolone.
* Patients presented with cutaneous rash during the 2 weeks prior to study initiation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2011-01; Primary Completion 2017-01 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Number of patients developing grade 2 / above rash under preventative treatment with ointment threolone, compared to the other 2 treatment arms. | 3 years

SECONDARY OUTCOMES:
Number of patients developing a rash under preventative treatment with ointment threolone, compared to the other 2 treatment arms | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Davidoff Center, Rabin Medical Center, Beilinson, Petah Tikva, Israel, Israel

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Lee JE, Lee SJ, Lee HJ, Lee JH, Lee KH. Severe acneiform eruption induced by cetuximab (Erbitux). Yonsei Med J. 2008 Oct 31;49(5):851-2. doi: 10.3349/ymj.2008.49.5.851. PMID 18972607
- [Background] Lacouture ME, Mitchell EP, Piperdi B, Pillai MV, Shearer H, Iannotti N, Xu F, Yassine M. Skin toxicity evaluation protocol with panitumumab (STEPP), a phase II, open-label, randomized trial evaluating the impact of a pre-Emptive Skin treatment regimen on skin toxicities and quality of life in patients with metastatic colorectal cancer. J Clin Oncol. 2010 Mar 10;28(8):1351-7. doi: 10.1200/JCO.2008.21.7828. Epub 2010 Feb 8. PMID 20142600